CLINICAL TRIAL: NCT01610401
Title: Can Metformin Prevent Endothelial Ischemia and Reperfusion Injury? The Metformin-FMD Trial
Brief Title: The Metformin-FMD Trial
Acronym: MetFMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Metformin-FMD 001
Record Dates: First submitted 2012-05-25; First posted 2012-06-04 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2012-02

CONDITIONS: Ischemia Reperfusion Injury; Endothelial Function
MeSH Terms: conditions — Reperfusion Injury | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pretreatment with metformin (Active Comparator): Pretreatment with metformin 500 mg three times a day for 3 days.
  Interventions: Drug: Metformin
- No pretreatment. (No Intervention): no intervention
- Pretreatment with Metformin/caffeine (Active Comparator): to study whether caffeine (4 mg/kg intravenously over 10 minutes) attenuates the protective effect of metformin (500 mg three times a day for 3 days) on FMD after ischemia/reperfusion
  Interventions: Drug: Pretreatment with metformin in combination of infusion of caffeine.
- No metformin, only pretreatment with caffeine (Other): No pretreatment with metformin, FMD measurement after forearm ischemia/reperfusion and infusion of caffeine (4 mg/kg intravenously over 10 minutes).
  Interventions: Drug: No pretreatment with metformin in combination with infusion of caffeine

INTERVENTIONS:
Drug: Metformin — metformin 500 mg three times a day, for 3 days
  Arms: Pretreatment with metformin
Drug: Pretreatment with metformin in combination of infusion of caffeine. — Pretreatment with metformin 500 mg three times a day for 3 days, in combination with pretreatment with caffeine (4 mg/kg intravenously over 10 minutes) prior to FMD measurement
  Arms: Pretreatment with Metformin/caffeine
Drug: No pretreatment with metformin in combination with infusion of caffeine — No pretreatment with metformin in combination with pretreatment with caffeine (4 mg/kg intravenously over 10 minutes).
  Arms: No metformin, only pretreatment with caffeine

SUMMARY:
In acute myocardial infarction early restoration of coronary blood flow is the most effective strategy to limit infarct-size. Paradoxically, reperfusion itself also aggravates myocardial injury and contributes to final infarct size, a process termed 'reperfusion injury'. Ischemia and reperfusion (IR)-induced endothelial dysfunction seems to play a pivotal role in this process, resulting in vasoconstriction and reduced blood flow to the already ischemic tissue. Recently, it has been shown that the glucose-lowering drug metformin is able to limit IR-injury in murine models of myocardial infarction, probably by increased formation of the endogenous nucleoside adenosine. In the current research proposal, the investigators aim to translate this finding to the human in vivo situation, using flow-mediated dilation (FMD) of the brachial artery as a well-validated model of (endothelial) IR-injury.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-50 years
* Written informed consent

Exclusion Criteria:

* Smoking
* Hypertension (in supine position: systolic BP > 140 mmHg, diastolic BP > 90 mmHg)
* Hyperlipidaemia (fasting total cholesterol > 5.5 mmol/L or random > 6.5 mmol/L)
* Diabetes Mellitus (fasting glucose > 7.0 mmol/L or random glucose > 11.0 mmol/L)
* History of any cardiovascular disease
* Concomitant use of medication
* Renal dysfunction (MDRD < 60 ml/min)
* Professional athletes

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Metformin-FMD trial: The effect of pretreatment with metformin on FMD of the brachial artery after forearm ischemia and reperfusion. | approx. 6 months
  Metformin-FMD trial: To study the effect of oral pretreatment with metformin (500 mg three times ad ay for 3 days) on flow mediated dilation of the brachial artery after 20 minutes of forearm ischemia and 20 minutes of reperfusion in healthy volunteers.
Control trial: the effect of caffeine on the protective effect of metformin on FMD after ischemia and reperfusion. | approx. 6 months
  Control trial: when metformin displays a protective effect on endothelial function, we will conduct a second experiment to study whether caffeine, an adenosine receptor antagonist, attenuates the protective effect of metformin on flow mediated dilation after 20 minutes of ischemia and 20 minutes of reperfusion in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: N. Riksen, MD, PhD, Principal Investigator — Radboud University Medical Center; G.A. Rongen, M.D., Principal Investigator — Radboud University Medical Center; D.H. Thijssen, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] El Messaoudi S, Schreuder TH, Kengen RD, Rongen GA, van den Broek PH, Thijssen DH, Riksen NP. Impact of metformin on endothelial ischemia-reperfusion injury in humans in vivo: a prospective randomized open, blinded-endpoint study. PLoS One. 2014 Apr 22;9(4):e96062. doi: 10.1371/journal.pone.0096062. eCollection 2014. PMID 24755906